CLINICAL TRIAL: NCT05366920
Title: Day-care Laparoscopic Cholecystectomy With Diathermy Hook Versus 5mm Suction Irrigation Blunt Dissection: a Randomized Study
Brief Title: Cholecystectomy Blunt Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Imam Mohammad ibn Saud Islamic University (Other)
Responsible Party: Principal Investigator, mohammad bukhetan alharbi, associate professor, Imam Mohammad ibn Saud Islamic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHOLECYSTECTOMY BLUNT
Record Dates: First submitted 2022-04-17; First posted 2022-05-09 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Cholecystolithiasis; Cholelithiasis; Gallstones; Biliary Tract Diseases; Digestive System Diseases; Gallbladder Diseases; Calculi; Pathological Conditions, Anatomical
MeSH Terms: conditions — Cholecystolithiasis; Cholelithiasis; Gallstones; Biliary Tract Diseases; Digestive System Diseases; Gallbladder Diseases; Calculi; Pathological Conditions, Anatomical | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional diathermy hook (Active Comparator): Laparoscopic cholecystectomy made with diathermy hook starting from Calot´s triangle Intervention: Procedure: dissection of gallbladder in laparoscopic cholecystectomy
  Interventions: Procedure: dissection of gallbladder in laparoscopic cholecystectomy
- 5 mm suction irrigation blunt dissection (Active Comparator): Laparoscopic cholecystectomy made with 5mm suction irrigation blunt dissection starting from gallbladder fundus Intervention: Procedure: dissection of gallbladder in laparoscopic cholecystectomy
  Interventions: Procedure: dissection of gallbladder in laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: dissection of gallbladder in laparoscopic cholecystectomy — Laparoscopic cholecystectomy with diathermy hook starting from triangle of Calot
Procedure: dissection of gallbladder in laparoscopic cholecystectomy — laparoscopic cholecystectomy with 5mm suction irrigation blunt dissection starting from fundus

SUMMARY:
Day case laparoscopic cholecystectomy can be made with conventional diathermy hook starting at triangle of Calot´s. 5mm suction irrigation blunt dissection starting from the gallbladder fundus is another option. The aim is to test the hypothesis that with 5mm suction irrigation blunt dissection technique a better same day discharge and a shorter operative time can be achieved.

DETAILED DESCRIPTION:
After initiation of general anaesthesia patients are randomized either to conventional(cautery) or 5mm suction irrigation blunt dissection group. The patients and recovery room personnel are blinded to the operative technique used.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* BMI under 35
* normal liver enzymes
* no bile duct dilatation in ultrasound
* cholecystolithiasis

Exclusion Criteria:

* NSAID allergy
* previous upper gi-surgery
* common bile duct stones in preoperative imaging
* history of severe acute pancreatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
number of days for discharge after surgery | 30 days
operative time | 30 days
intraoperative bleeding amount | 30 days
  bleeding which require suction or draining

SECONDARY OUTCOMES:
type of analgesic and dose | 30 days
number of events of postoperative nausea and vomiting which require anti emetic drug | 30 day
number of days after surgery when readmission is required | 30 days
presence of a morbidity | 30days
  number of days needed for discharge from service

CONTACTS AND LOCATIONS:
Locations (1):
- Central fourth Health Cluster, Hail, Saudi Arabia